CLINICAL TRIAL: NCT06795763
Title: Chronic Total Occlusion (CTO) Crossing, Re-entry and Imaging With the Acolyte™ Catheter System in Subjects Undergoing Percutaneous Coronary Interventional (PCI) Procedures
Brief Title: Acolyte CTO-PCI Study: Imaging and Catheter System to Treat Patients With Coronary Chronic Total Occlusion, Who Have Persistent Symptoms Following Medical Therapy and Are Undergoing Percutaneous Coronary Interventional Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Simpson Interventions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP24001
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Coronary Chronic Total Occlusions; Ischemic Heart Disease; Ischemic Heart Disease (IHD); Ischemic Heart Disease Chronic
Keywords: CTO-PCI; CTO
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CTO-PCI Procedure with Acolyte Catheter System (Experimental)
  Interventions: Device: CTO-PCI Procedure with Acolyte Catheter System

INTERVENTIONS:
Device: CTO-PCI Procedure with Acolyte Catheter System — Acolyte Catheter System is used to facilitate placement and positioning of guidewires and catheters within the coronary vasculature for the treatment of patients with coronary chronic total occlusions with persistent symptoms following medical therapy. The device provides real-time visualization of a coronary chronic total occlusion allowing for guidewire placement in the true lumen of the target vessel and subsequent revascularization.

SUMMARY:
This is a study to evaluate the safety and effectiveness of the Acolyte Catheter System used in CTO-PCI procedures. The system will be used for the placement and positioning of guidewires and catheters in the coronary vasculature for the treatment of patients with coronary chronic total occlusions with persistent symptoms following medical therapy.

DETAILED DESCRIPTION:
This is a study to evaluate the safety and effectiveness of the Acolyte™ Catheter System used in CTO-PCI procedures as follows:

* Evaluate angiographic confirmation of guidewire placement beyond the CTO, in the true vessel lumen, in which the investigational device was utilized to facilitate crossing and/or re-entry.
* Evaluate in-hospital major adverse cardiac events (MACE).

Acolyte™ Optical Coherence Tomography (OCT) imaging will be utilized in all cases to inform guidewire advancement in the direction of true lumen. Additionally, Acolyte™ OCT imaging will be used to guide re-entry from the subintimal space to the true lumen.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age at the time of consent
* Subject is on medical therapy and continues to experience clinical symptoms considered suggestive of ischemic heart disease (e.g., chest pain or discomfort, heart failure) or has evidence of myocardial ischemia (e.g., abnormal functional study) attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization
* Female subjects of reproductive potential must have a negative pregnancy test per standard of care for PCI
* Subject is willing and able to provided written informed consent
* Subject is willing to and able to comply with the study protocol requirements including all follow up visits post-procedure

Exclusion Criteria:

* Subject has history of allergy to iodinated contrast that cannot be managed medically
* Subject has evidence of acute myocardial infarction (MI) within 72 hours prior to the intended treatment
* Subject has had previous coronary interventional procedure of any kind within 30 days prior to the investigational procedure
* Atherectomy procedure is planned for the target lesion
* History of stroke or transient ischemic attack within 6 months prior to procedure
* Active peptic ulcer or upper gastrointestinal bleeding within 6 months prior to procedure
* History of bleeding diathesis or coagulopathy or refusal of blood transfusions
* Other pathology such as cancer, known mental illness, etc., or other condition which might, in the opinion of the Investigator, put the patient at risk or confound the results of the study
* Subject participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with this study's endpoints; or requires coronary angiography, intravascular ultrasound, or other coronary artery imaging procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Procedure Success - Visualization of Guidewire | From the beginning of the study procedure to the end of the study procedure
  Procedure success is defined as angiographic visualization of a guidewire facilitated by the Acolyte Catheter System, in a distal position of the CTO in the true lumen of the vessel.
Procedure Success - Absence of Major Adverse Cardiac Events | From the beginning of the study procedure until discharge or 24 hours after the procedure (whichever comes first)
  Absence of in-hospital major adverse cardiac events (MACE). MACE is defined as any serious adverse experience that includes cardiac death, target lesion revascularization, or post-procedural myocardial infarction (with CK-MB >= 10x URL or >= 5x URL with new pathological Q waves in >= 2 contiguous leads or new persistent left bundle branch block (LBBB)).

SECONDARY OUTCOMES:
Successful Recanalization | From the beginning of the study procedure to the end of the study procedure
  Frequency of successful recanalization defined as angiographic confirmation of crossing the chronic total occlusion and restoring blood flow to the affected area
In-Hospital: Frequency of Major Adverse Cardiac Events (MACE) | From the beginning of the study procedure until discharge or 24 hours after the procedure (whichever comes first)
  Any serious adverse experience that includes cardiac death, target lesion revascularization, or post-procedural myocardial infarction.
30-Day: Frequency of Major Adverse Cardiac Events (MACE) | 30 Day Follow-up
  Any serious adverse experience that includes cardiac death, target lesion revascularization, or post-procedural myocardial infarction.
Safety - Blood Vessel Perforation | From the beginning of the study procedure to the end of the study procedure
  Frequency of clinically significant perforation (perforation that results in hemodynamic instability and/or requiring intervention including pericardiocentesis, embolization, prolonged balloon occlusion, stent graft, or comparable therapy).
Procedure: Serious Adverse Events Related to Study Device or Procedure | From the beginning of the study procedure until discharge or 24 hours after the procedure (whichever comes first)
  Frequency of serious adverse events (SAEs) related to the study device or procedure
30-Day: Serious Adverse Events Related to Study Device or Procedure | 30 Day Follow-up
  Frequency of serious adverse events (SAEs) related to the study device or procedure
3-Month: Serious Adverse Events Related to Study Device or Procedure | 3-Month Follow-up
  Frequency of serious adverse events (SAEs) related to the study device or procedure
Procedure: Non-serious Adverse Events Related to Study Device or Procedure | From the beginning of the study procedure until discharge or 24 hours after the procedure (whichever comes first)
  Frequency of non-serious adverse events related to the study device or procedure
30-Day: Non-serious Adverse Events Related to Study Device or Procedure | 30 Day Follow-up
  Frequency of non-serious adverse events related to the study device or procedure
Procedure: Time for Guidewire to Cross Chronic Total Occlusion (CTO) | From the beginning of the study procedure to the end of the study procedure
  Time from initial CTO guidewire entered into guide to guidewire crossing chronic total occlusion
Procedure: Fluoroscopy Time | From the beginning of the study procedure to the end of the study procedure
  Total fluoroscopy time during procedure
Procedure: Technical Success | From the beginning of the study procedure to the end of the study procedure
  Crossing chronic total occlusion and/or re-entry success
Change from Baseline in Seattle Angina Questionnaire-7 at 30 Days | Baseline and 30 Days
  Change from Baseline in Mean Seattle Angina Questionnaire-7 at 30 Days
Change from Baseline in Seattle Angina Questionnaire-7 at 3 Months | Baseline and 3 Months
  Change from Baseline in Mean Seattle Angina Questionnaire-7 at 3 Months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NCH Healthcare System, Naples, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St. Francis Hospital, Roslyn, New York
  - PharmaTex Research, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: No